A prospective, double-masked, randomized, multi-center, active-controlled, parallel-group, 3-month study assessing the safety and ocular hypotensive efficacy of PG324 Ophthalmic Solution compared to AR-13324 Ophthalmic Solution 0.02% and latanoprost ophthalmic solution 0.005% in subjects with elevated intraocular pressure

NCT02674854

30January2017

# STATISTICAL ANALYSIS PLAN Version 1.0 30 December

A prospective, double-masked, randomized, multi-center, active-controlled, parallel-group, 3-month study assessing the safety and ocular hypotensive efficacy of PG324 Ophthalmic Solution compared to AR-13324 Ophthalmic Solution 0.02% and latanoprost ophthalmic solution 0.005% in subjects with elevated intraocular pressure

#### PROTOCOL NUMBER PG324-CS302

#### SPONSORED BY

Aerie Pharmaceuticals, Inc. 135 US Highway 206, Suite 15 Bedminster, NJ 07921 Telephone: (908) 470-4320 Fax: (908) 325-0266

#### PREPARED BY



This document contains Aerie Pharmaceuticals, Inc. (Aerie) information that is confidential, a trade secret and/or proprietary in nature. It is loaned to you for your confidential use on behalf of Aerie and is not to be photocopied, disclosed or transmitted to any other person or party who is not covered by a Confidential Disclosure Agreement with Aerie.

Version 1.0 

# **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|----------------|-------------------|------------------|
| 0.1 | December 16, 2016 | Draft |
| 1.0 | January 30, 2017 | Final |




# TABLE OF CONTENTS

| LIS | T OF | ABBREVIATIONS | 6 |
|---|---|---|---|
| 1. | PUR | RPOSE OF THE ANALYSES | 7 |
| 2. | PRC | OTOCOL SUMMARY | 8 |
| | 2.1<br>2.2<br>2.3<br>2.4<br>2.5 | Study Objectives Overall Study Design and Plan Study Population Treatment Regimens Treatment Group Assignments or Randomization Sample Size Determination | 8<br>11<br>11 |
| 3. | GEN | NERAL ANALYSIS AND REPORTING CONVENTIONS | 13 |
| 4. | ANA | ALYSIS POPULATIONS | 14 |
| | 4.2<br>4.3 | Randomized Population Intent-to-Treat Population (ITT) Per-protocol Population (PP) Safety Population | 14<br>14 |
| <b>5.</b> | STU | DY SUBJECTS | 15 |
| | | Disposition of Subjects | |
| 6. | | MOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| | 6.2 | Demographics and Baseline Characteristics | 16 |
| 7. | MEA | ASUREMENTS OF TREATMENT COMPLIANCE | 18 |
| 8. | EFF | TICACY EVALUATION | 19 |
| | 8.1<br>8.2<br>8.3 | Overview of Efficacy Analysis Issues. 8.1.1 Handling of Dropouts or Missing Data. 8.1.2 Multicenter Studies. 8.1.3 Assessment Time Windows. Efficacy Variables and Primary Hypotheses. Analysis Methods. 8.3.1 Primary Efficacy Analyses. 8.3.2 Secondary Efficacy Analyses. | 19 19 19 19 19 21 22 24 |
| | | Examination of Subgroups | |
| 9. | | ETY EVALUATION | |
| | 9.2<br>9.3<br>9.4<br>9.5<br>9.6 | Overview of Safety Analysis Methods. Extent of Exposure | 26<br>27<br>27<br>28<br>28 |
| | | 9.6.3 Visual Acuity | |

| | 9.6.4 | Dilated Ophthalmoscopy and Cup-to-Disc Ratio | 28 |
|-----|---------|------------------------------------------------------|----|
| | 9.6.5 | | |
| | 9.6.6 | | 29 |
| | 9.6.7 | Pupil Size | |
| | 9.6.8 | _ | |
| | 9.6.9 | Visual Field Examination, Pachymetry, and Gonioscopy | |
| 10. | PHARMA | COKINETIC EVALUATION | 31 |
| 11. | OTHER A | NALYSES | 32 |
| 12. | INTERIM | ANALYSES AND DATA MONITORING | 33 |
| 13. | CHANGES | S TO THE ANALYSES PLANNED IN THE PROTOCOL | 34 |
| 14. | REFEREN | ICES | 35 |
| 15. | APPENDI | CES | 36 |
| 16. | ATTACH | MENTS | 38 |

#### LIST OF ABBREVIATIONS

AE Adverse Event

ANCOVA Analysis of Covariance ANOVA Analysis of Variance

AR-13324 AR-13324 (Netarsudil Ophthalmic Solution) 0.02%

BCVA Best Corrected Visual Acuity

CRF Case Report Form
CSR Clinical Study Report

ETDRS Early Treatment of Diabetic Retinopathy Study

ICF Informed Consent Form

ICH International Conference on Harmonization

IOP Intraocular Pressure

LOCF Last Observation Carried Forward

logMAR Logarithm of the Minimum Angle of Resolution

LS Mean Least Squares Mean

ITT Intent-to-treat

IWRS Interactive Web Response System MMRM Mixed Model Repeated Measures

OAG Open-Angle Glaucoma
OHT Ocular Hypertension

OU Both eyes
PP Per-Protocol
QD Once-daily

SAE Serious Adverse Event SAP Statistical Analysis Plan SAS Statistical Analysis Software

SD Standard Deviation

SE Standard Error

TEAE Treatment Emergent Adverse Event

VF Visual Fields


## 1. PURPOSE OF THE ANALYSES

This statistical analysis plan (SAP) is being developed after review of the Aerie Pharmaceuticals, Inc., protocol number PG324-CS302 (Amendment 1, dated 22 December 2015) but before any analyses of the data. The SAP contains detailed information to aid in the performance of the statistical analysis and reporting of the study data for use in the final clinical study report (CSR). This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed and will be identified in the CSR.


#### 2. PROTOCOL SUMMARY

# 2.1 Study Objectives

The primary objectives of this study are to evaluate:

- The ocular hypotensive efficacy of PG324 Ophthalmic Solution, QD relative to each of its active components, AR-13324 0.02% (ie. Netarsudil 0.02%), QD and Latanoprost 0.005%, QD over a 3-Month period
- The ocular and systemic safety of PG324 Ophthalmic Solution over a 3-month period relative to each of its active components, Netarsudil 0.02% and latanoprost 0.005%, over a 3-month period

The secondary objectives of this study are to evaluate:

- Mean intraocular pressure (IOP) within a treatment group at each post-treatment time point
- Mean diurnal IOP within a treatment group at each post-treatment visit
- Mean change from diurnally adjusted baseline IOP at each post-treatment time point
- Mean change from baseline in diurnal IOP at each post-treatment visit
- Mean percent change from diurnally adjusted baseline IOP at each post-treatment time point
- Mean percent change from baseline in diurnal IOP at each post-treatment visit
- Percentages of subjects achieving pre-specified mean, mean change, and percent mean change in diurnal IOP levels

# 2.2 Overall Study Design and Plan

This is a 3-month, double-masked, randomized, multi-center, active-controlled, parallel-group safety and efficacy trial for reduction of elevated intraocular pressure (IOP) with PG324 Ophthalmic Solution compared to each of its active components, AR-13324 0.02% and latanoprost 0.005%, in subjects at least 18 years of age (at least 19 years for subjects in Canada) with open angle glaucoma (OAG) or ocular hypertension (OHT). All investigational products will be dosed QD (PM). Eligible subjects are required to have a diagnosis of either OAG or OHT in both eyes. Subjects who agree to participate in this study and are randomized in the study will attend a total of 6 study visits: a Screening Visit, Qualification Visit #1, Qualification Visit #2/Day 1 (baseline), Week 2 (Day 15), Week 6 (Day 43), and Month 3 (Day 90). Subjects currently using ocular hypotensive medication will be required to undergo a wash out for a specified period (5 days-4 weeks, depending on the medication) prior to attending Qualification Visit #1. Subjects eligible to be enrolled in this study must meet all inclusion criteria and none of the exclusion criteria at each of the Screening Visit and Qualification Visits #1 and #2. Among multiple procedures, subjects will receive an eye examination including IOP measurements at Oualification Visits #1 and #2 and, if deemed eligible, will be enrolled at Oualification Visit #2 and assigned to 1 of 3 investigational products in a 1:1:1 ratio according to a computer-generated randomization list. Approximately 690 subjects will be randomized in this study.

Randomization will take place using IWRS methodology and will stratify subjects by site and by maximum baseline IOP ( $< 25 \text{ mmHg vs} \ge 25 \text{ mmHg}$ ). Randomized subjects will dose the


assigned investigational product in both eyes QD in the evening beginning on Day 1 and up to and including the evening prior to the Month 3 visit.

Procedures conducted at each visit will include safety and efficacy measurements, including IOP at the following time points: 08:00, 10:00, and 16:00 hours. Subjects will be seen in the clinic for safety and efficacy assessments during the treatment period at Weeks 2 and 6, and Month 3. Following completion of the Month 3 study visit procedures, subjects will exit from the study. For subjects who discontinue early, every possible effort will be made to assure there is an exit visit that includes all required examinations listed for Visit 6 (Month 3) and dilated ophthalmoscopy.

At Screening (Visit 1), an examination will be conducted, including measurements of heart rate and blood pressure (vital signs), urine pregnancy test (for women of child bearing potential), and an ophthalmic examination (to include ocular symptoms, best corrected visual acuity (BCVA), central corneal thickness by ultrasound pachymetry (may be taken within 1 week of Visit 1), intraocular pressure (IOP; before pupil dilation), biomicroscopy, specular microscopy, and dilated ophthalmoscopy). Visual fields and gonioscopy may be taken up to three months prior to randomization (Visit 3). Subject symptoms will be queried and blood samples will be taken for clinical chemistry and hematology. All individuals who are qualified for enrollment will have their current ocular hypotensive therapy reviewed to determine the appropriate washout period, prior to Visit 2, as specified in Section 5.7.1 of the protocol.

At Visit 2 (Qualification #1, Day -2 to -7, 08:00 hours), potential study subjects will again be questioned with respect to changes in their health (to be recorded as medical history) and concomitant medication use. Study inclusion/exclusion criteria will be reassessed to confirm eligibility. BCVA, vital signs, IOP, and biomicroscopy assessments will again be performed. The potential subject must have a post-washout IOP > 20 mmHg and < 36 mmHg in both eyes to qualify for further participation. This is the first of four qualifying IOPs for randomization

Qualified subjects will return for Visit 3 (Qualification #2, Baseline, Day 1) 2 to 7 days after Visit 2 at 3 time points. At Visit 3.0 (08:00 hours), testing will include recording symptomatology, vital signs, BCVA, IOP, biomicroscopy, and pupil size assessments. Any symptoms reported at this visit should be entered into medical history. The potential subject must have a post-washout IOP > 20 mmHg and < 36 mmHg in both eyes to qualify for further participation. This is the second of four qualifying IOPs for randomization.

Qualifying subjects will return for two additional visits on this day (Visit 3.1 at 10:00 hours and Visit 3.2 at 16:00 hours) during which symptomatology, IOP, and biomicroscopy assessments will be performed. The subject must have an IOP of > 17 mmHg and < 36 mmHg in both eyes to continue to be qualified. These are the third and the fourth of four qualifying IOPs for randomization.

In summary, the following IOP criteria must be met at the qualifying visits in both eyes for the subject to qualify for the study:

| IOP Requirement |
|-----------------|
| 1 |


| | (mmHg) |
|-------------------------------|-------------|
| Visit 2, Day-2 to -7, 8:00 | > 20 & < 36 |
| hours | |
| Visit 3.0, Day 1, 8:00 hours | > 20 & < 36 |
| Visit 3.1, Day 1, 10:00 hours | > 17 & < 36 |
| Visit 3.2, Day 1, 16:00 hours | > 17 & < 36 |

Subjects qualify in both eyes based upon IOP and ocular history.

For each qualification visit, individuals who don't meet the IOP requirement may return for up to 2 additional unscheduled qualification visits within 1 week of failing the specific qualification visit. Individuals returning at an unscheduled visit within 1 week are required to only re-measure IOP in both eyes. Upon return, such individuals would need to qualify at 08:00, 10:00 and 16:00 hours to continue the study.

For a subject who qualifies, the study eye will be the eye with the higher IOP at 08:00 hours on Visit 3. If both eyes have the same IOP at 08:00 hours on Visit 3, then the right eye will be the study eye. In each subject, both eyes will be treated.

At this point, eligible subjects will be enrolled and assigned to an investigational product through an IWRS system according to a computer-generated randomization list. The first kit removed from an investigational product packer assigned through the IWRS system to the eligible subject will be dispensed unopened to the subject, along with written storage instructions.

# Subjects will be:

• Instructed to self-administer their masked medication at home between 20:00-22:00 hours (8 PM - 10 PM) beginning with the evening dose on that day

Subjects will return for post-treatment Visits 4.0, 4.1, and 4.2 (Week 2 [Day 15]; 08:00, 10:00, and 16:00 hours), Visits 5.0, 5.1, and 5.2 (Week 6 [Day 43]; 08:00, 10:00, and 16:00 hours), and Visits 6.0, 6.1, and 6.2 (Month 3 [Day 90]; 08:00, 10:00, and 16:00 hours). Symptomatology and non-dilated eye examinations including IOP and biomicroscopy will be conducted at all of these visits. Vital signs, comfort test, and BCVA will also be conducted at the 08:00 hour visits. Any symptoms reported, or clinical signs observed which have worsened, either from baseline or from previous visits at these post-dose visits, will be recorded as treatment emergent adverse events (TEAEs).

• Other tests will be performed in addition to those mentioned in the previous paragraph: At Visit 6.0 (Month 3 [Day 90], 08:00 hours), a urine pregnancy test will be performed, and visual fields, specular microscopy, pachymetry, and pupil size will be measured. Blood will be drawn for clinical chemistry and hematology labs as well. A dilated ophthalmoscopy will be performed at Visit 6.2 (Month 3 [Day 90], 16:00 hours), with an exemption that a dilated ophthalmoscopy at Visit 6.0 at 08:00 hours should be performed for all non-completing subjects during the exit visit.


A study schedule of events table is presented in Appendix 1.

# 2.3 Study Population

The study population includes subjects aged 18 years or older (at least 19 years for subjects in Canada) with a diagnosis of OAG or OHT. Subjects must have an unmedicated (post-washout) IOP > 20 and < 36 mmHg at 2 eligibility visits (08:00 hour), 2-7 days apart and > 17 and < 36 mmHg at 10:00 and 16:00 hours at the second qualification visit in both eyes. Corrected visual acuity in each eye must be +1.0 logMAR or better by early treatment of diabetic retinopathy study (ETDRS). The subject must also be willing to give signed inform consent and follow study instructions. The specific inclusion and exclusion criteria can be found in Sections 4.2 and 4.3 of the study protocol.

# 2.4 Treatment Regimens

There will be 3 treatments in this study:

- PG324 (Netarsudil 0.02% and latanoprost 0.005%) Ophthalmic Solution, QD
- Netarsudil Ophthalmic Solution 0.02%, QD
- Latanoprost Ophthalmic Solution 0.005%, QD

Each investigational product is being dosed QD OU (in the evening between 20:00 and 22:00 hours)

Subjects will be instructed to self-administer their masked medication once a day (QD) in the evening between 20:00-22:00 hours (8pm - 10pm). All treatments will be dosed in both eyes (OU). The treatment period will be 90 days.

## 2.5 Treatment Group Assignments or Randomization

A randomization code for allocating the treatments was prepared by an independent biostatistician, who was not involved in the day-to-day conduct of the study, and provided in confidence to the VP of Manufacturing at Aerie, the clinical supply company chosen by Aerie, and the Interactive Web Response (IWR) system personnel. At Visit 3.2 (Day 1), qualified subjects will be randomized in a 1:1:1 ratio to receive PG324 Ophthalmic Solution, Netarsudil Ophthalmic Solution 0.02%, or Latanoprost Ophthalmic Solution 0.005% (stratified by investigative site and by maximum baseline IOP [< 25 mmHg vs ≥ 25 mmHg]). Treatment assignments were masked to the Investigator, the Sponsor team members involved in the day-to-day oversight of the clinical study and employees of the CRO administrating the study for the Sponsor, and the study subjects. At the end of the study, the randomized treatment assignments will be presented in a data listing.

#### 2.6 Sample Size Determination

One-hundred ninety six (196) subjects per arm completing 3 months of treatment yields at least 90% power to conclude statistical superiority of PG324 to latanoprost and > 99% power to conclude statistical superiority of PG324 to Netarsudil at all nine time points assuming a two-sided alpha = 0.05, a true mean difference of 1.5 mmHg (to latanoprost) and 2.0 mmHg (to Netarsudil), a common standard deviation of 3.5 mmHg at each time point, and independence


among time points. Power increases as the correlation among time points increases. Therefore, 196 subjects per arm yields at least 90% power to conclude superiority to both controls over all nine time points.


# 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies may be given in the specific detailed sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

All continuous study assessments will be summarized by treatment and time point (as applicable) using descriptive statistics (n, mean, median, standard deviation (SD), minimum, and maximum). All categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and percentages.

All study data will be listed by treatment, subject, visit, and time point (as applicable).

Hypothesis testing, unless otherwise indicated, will be performed at a 2-sided 0.05 significance level. When applicable, two-sided 95% confidence intervals will be reported. All p-values will be displayed to four decimal places, with p-values less than 0.0001 presented as '<0.0001' and p-values greater than 0.9999 presented as '>0.9999'. Differences between PG324 and each comparator (latanoprost and Netarsudil) will be calculated as PG324 – comparator.

For diurnally adjusted IOP, baseline will refer to the time-relevant measure at Visits 3.0 through 3.2 (e.g. IOP at 08:00 hours at Visit 3.0 will be the baseline for 08:00 hours at Visits 4.0, 5.0, and 6.0, etc.; IOP at 10:00 hours at Visit 3.1 will be the baseline for 10:00 hours at Visits 4.1, 5.1, and 6.1, etc.). For mean diurnal IOP, baseline will refer to the mean diurnal IOP at Visit 3. For all other variables, baseline is defined as the last measurement prior to the first dose of study medication. Change from baseline will be calculated as follow-up visit – baseline visit.

All study data will be listed by subject, treatment, and time point (as applicable). In the listings, individual subjects will be identified by a combination of site number and subject number, e.g., XXX-YYY, where XXX is the site number and YYY is the subject number.

All data analysis will be performed by after the study is completed and the database has been locked and released for un-masking. Statistical programming and analyses will be performed using SAS® Version 9.4. Output will be provided in rtf format for tables and pdf format for tables, listings, and figures.


#### 4. ANALYSIS POPULATIONS

# 4.1 Randomized Population

The randomized population will include all subjects who were randomized to treatment. Baseline variables and demographic characteristics will be summarized for this population.

# 4.2 Intent-to-Treat Population (ITT)

The ITT population will include all randomized subjects who have received at least one dose of study medication. This population will be the primary population for efficacy analyses and will be used to summarize all efficacy variables and will summarize subjects as randomized.

# 4.3 Per-protocol Population (PP)

The PP population is a subset of the ITT population, which will include those subjects (and their visits) who do not have major protocol violations likely to seriously affect the primary outcome of the study as judged by a masked evaluation prior to the unmasking of the study treatment. This population will be the secondary population for efficacy analyses and will be used to summarize a subset of efficacy variables. If the PP and ITT populations are exactly the same, then additional efficacy analyses on the PP population will not be performed. The PP population will summarize subjects as treated.

# 4.4 Safety Population

The safety population will include all randomized subjects who have received at least one dose of study medication. This population will be used to summarize safety variables and will summarize subjects as treated.


## 5. STUDY SUBJECTS

# 5.1 Disposition of Subjects

Subject randomization, analysis populations, study completion, and withdrawal from the study will be summarized and listed for all randomized subjects. The summary table will include the numbers of subjects randomized and included in the analysis populations by randomized treatment group for the ITT population and by actual treatment group for the PP and Safety populations. It will also include the numbers of subjects who completed and discontinued from the study. The reasons for subject discontinuation and test agent discontinuation will be summarized for the applicable subjects. Reasons for subject discontinuation will include adverse event (AE), withdrawal of consent, non-compliance, lost to follow-up, lack of efficacy, disallowed concurrent medication, investigator decision, protocol violation, death, and an "other" category for reasons other than those previously listed.

By-subject listings will include randomization information, actual treatment assigned, first and last dose dates, exposure, study eye, and analysis population inclusion. For subjects who prematurely discontinue following randomization, an additional by-subject listing will be provided that shows treatment assignment, gender, age, date of last visit, date of last dose, treatment duration at time of discontinuation, study day of discontinuation, and reason for discontinuation. Study day of discontinuation will be calculated as (date of discontinuation – date of Visit 3 date +1). Note that date of first dose is not collected, but will be assumed to be the Visit 3 date. Treatment duration will be calculated as the (Date of Last Dose – Visit 3 Date + 1).

#### **5.2** Protocol Deviations

Protocol deviations will be evaluated for all subjects in the safety population. Major protocol violations will be judged by a masked evaluation and summarized in writing prior to the unmasking of the study treatment, for the purpose of selecting the PP population. All subjects having a protocol deviation will be identified in a subject data listing. The number of subjects with protocol deviations and level of deviations (major or minor) will be summarized by treatment group and severity of the deviation along with the disposition data.

Concomitant medications used during the study will be reviewed by study staff to identify deviations associated with the use of prohibited medications during the double-masked treatment period. Procedural deviations will be determined from administrative requirements and any other comments recorded on the CRF or supporting documentation.

Failure to meet all Protocol Inclusion Criteria or meeting any Exclusion Criterion will also be considered for categorization as a major Protocol Deviation. Inclusion and Exclusion Criteria will be presented in a by-subject listing.


#### 6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

# 6.1 Demographics and Baseline Characteristics

Demographic and baseline characteristics will be summarized by treatment group and listed for the randomized population. Demographic parameters will include gender, iris color, age in years at signing of informed consent form (ICF), race, ethnicity, prior hypotensive therapy, and time on current hypotensive therapy. Baseline characteristics will include study eye diagnosis of OHT or OAG, length of time since study eye diagnosis of OHT or OAG, study eye IOP at screening, and study eye mean diurnal IOP at baseline. Additionally, means for both the study eye and the fellow eye will be summarized separately for the baseline ocular measurements of deviation in visual fields, central corneal thickness, and cup to disc ratio.

Age will be reported in years and calculated in SAS using the formula:

$$Age = Floor ((ICFDT - DOB) / 365.25)$$

where ICFDT is the date the subject signed the informed consent, DOB is the subject's date of birth, and Floor takes the integer part of the result.

Tests of differences between the treatment groups will be performed for both demographic and baseline characteristics. Categorical responses will be tested using Fisher's exact tests. Continuous measures will be tested using an analysis of variance model with treatment as the only explanatory variable.

#### 6.2 Prior and Concomitant Medications

All medications which the subject has taken within 30 days prior to randomization and during the study will be recorded on the CRF. The name of the drug, dose, route of administration, duration of treatment, and indication will be recorded for each medication. For combination products (e.g., Contac®), the brand name is required. For non-combination products, the generic name is desired. The use of routine ophthalmic diagnostic pharmaceutical agents (e.g., fluorescein and local anesthetic) will be allowed, and individual documentation not required. Any change in dosing parameters should also be recorded on the CRF.

All prior and concomitant medications will be coded to preferred drug names and therapeutic drug class using the *WHO Drug Dictionary Enhanced* (2016, Q1 version). Use of concomitant medications will be summarized for each therapeutic drug class and each preferred drug name by treatment group. Subjects will be counted only once under each therapeutic drug class and preferred term for which they have used at least one concomitant medication. All prior and concomitant medication data will also be listed.

The class of prior hypotensive therapy, summarized on the baseline characteristic table and listed on the washout medication listing, will also be derived from the coded medication data. Classes include the following: Prostaglandins,  $\beta$ -adrenoceptor antagonists, adrenergic agonists (including  $\alpha$ -agonists such as brimonidine and apraclonidine), Muscarinic agonists (e.g., pilocarpine), and Carbonic anhydrase inhibitors (topical or oral). For the summary table, categories will be: combination therapy, prostaglandins (monotherapy), other (monotherapy), and no prior therapy.


Additionally, the following two classes will be summarized: prior prostaglandin therapy and no prior prostaglandin therapy.

# 6.3 Medical and Ocular History

A medical and ocular history will be collected at screening, including diagnosis, start date, and stop date (as applicable) or ongoing. For ocular history, the applicable eye(s) will be noted. Any change in the individual's baseline health status that occur after screening and prior to first dose of study medication should be reported as medical history events.

Ocular surgery and laser procedures will also be collected at screening including the procedure description, procedure date, and affected eye(s).

All medical history and ocular surgery/laser procedures data will be presented in a by-subject listing. Medical and ocular history will be coded to preferred terms and system organ class using the MedDRA Dictionary (Version: 19.0). Medical and ocular histories will be summarized for each system organ class and each preferred term by treatment group. Subjects will be counted only once under each system organ class and preferred term for which they have at least one medical/ocular history.

Study eye diagnosis will be derived from the coded ocular history data. The preferred terms of "Ocular hypertension" and "Open angle glaucoma" will be matched to the study eye selection page of the CRF. Analyses based on study diagnosis will use this definition.


# 7. MEASUREMENTS OF TREATMENT COMPLIANCE

All subjects will be instructed to follow once a day dosing regimen in the evening between 20:00 – 22:00 hours (8pm - 10pm). All treatments will be dosed in both eyes (OU).


## 8. EFFICACY EVALUATION

# 8.1 Overview of Efficacy Analysis Issues

#### 8.1.1 Handling of Dropouts or Missing Data

Any missing, unused, or spurious data will be noted in the final statistical report. Analyses will be performed primarily on the intent to treat population with multiple imputation techniques (eg, Monte Carlo Markov Chain) used to impute missing data and secondarily using: observed data only, last observation carried forward (LOCF) where LOCF will be performed using time-relevant measures (i.e. from the same time point of the most recent visit with a non-missing value); and baseline observation carried forward (BOCF) using time-relevant measures to determine the robustness of results.

#### 8.1.2 Multicenter Studies

This study will have approximately 50 different sites enrolling and treating subjects. The homogeneity of treatment effect across investigative sites will be examined by a model containing the additional factors of investigative site and its interaction with treatment for the primary IOP efficacy endpoint.

#### **8.1.3** Assessment Time Windows

In general, it is intended that all safety and efficacy data (with some exceptions) will be summarized at each time point collected regardless of assessment time windows. Because subjects may have an early termination visit at any time or may have unscheduled visits, the following conventions will be implemented.

For all safety data, the visit date or start date (e.g., adverse events) will be used to calculate study day, defined as the number of days from the day of first dose. The day of first dose (Visit 3) is considered study day 1, so study day will be computed as (date of data – Visit 3 + 1). Study day will be presented in listings for medical history, concomitant medications, and adverse events.

In all by-visit safety assessments, end of study visits and early termination visits will be combined in order to present all data available for each subject; early termination visits will not be windowed into the nearest fitting study visit. Each subject will have one end of study visit. For efficacy outcomes, early termination data will not be combined with end of study visit information as the timing of the outcome measure is integral to the analysis. Instead, the efficacy outcome will be windowed into the nearest study visit, where each follow-up visit through Month 3 has  $a \pm 3$  day window.

# 8.2 Efficacy Variables and Primary Hypotheses

- 1. The primary efficacy outcome will be the comparison of PG324 Ophthalmic Solution relative to each of its active components (Netarsudil 0.02% and latanoprost 0.005%) for:
  - Mean IOP within a treatment group at 08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 study visits


- 2. Secondary efficacy endpoints will include the comparison of PG324 Ophthalmic Solution relative to each of its active components (Netarsudil 0.02% and latanoprost 0.005%) for:
  - Mean IOP within a treatment group at each post-treatment time point
  - Mean diurnal IOP within a treatment group at each post-treatment visit
  - Mean change from diurnally adjusted baseline IOP at each post-treatment time point
  - Mean change from baseline in diurnal IOP at each post-treatment visit
  - Mean percent change from diurnally adjusted baseline IOP at each post-treatment time point
  - Mean percent change from baseline in diurnal IOP at each post-treatment visit
  - Percentages of subjects achieving pre-specified mean, mean change, and percent mean change diurnal IOP levels at each post-treatment time point:
    - o Diurnal mean IOP of  $\leq 22, \leq 21, \leq 20, \leq 19, \leq 18, \leq 17, \leq 16, \leq 15, \leq 14$
    - o IOP reduction from baseline of ≥2, ≥4, ≥6, ≥8, ≥10, ≥12 (IOP reduction at a visit from baseline was calculated as IOP [baseline] IOP [visit], using mean [integral or non-integral] IOP values)
    - IOP percent reduction from baseline of ≥5, ≥10, ≥15, ≥20, ≥25, ≥30, ≥35, ≥40
       (IOP percent reduction at a visit from baseline was calculated as [IOP reduction from baseline / IOP (baseline)] \* 100%)
- 3. The primary hypotheses are:
  - $H_{01}$ : The difference between study eyes treated with PG324 Ophthalmic Solution and study eyes treated with latanoprost Ophthalmic Solution 0.005% (PG324 latanoprost), in mean IOP at the following time points: 08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 Visits, is  $\geq$  0 mmHg for at least one time point over all visits
  - H<sub>11</sub>: The difference between study eyes treated with PG324 Ophthalmic Solution and study eyes treated with latanoprost Ophthalmic Solution 0.005% (PG324 latanoprost), in mean IOP at the following time points: 08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 Visits, is < 0 mmHg for all time points over all visits.
  - $H_{02}$ : The difference between study eyes treated with PG324 Ophthalmic Solution and study eyes treated with Netarsudil Ophthalmic Solution 0.02% (PG324 Netarsudil), in mean IOP at the following time points: 08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 Visits, is  $\geq 0$  mmHg for at least one time point over all visits.
  - H<sub>12</sub>: The difference between study eyes treated with PG324 Ophthalmic Solution and study eyes treated with Netarsudil Ophthalmic Solution 0.02% (PG324 Netarsudil), in mean IOP at the following time points: 08:00, 10:00, and 16:00 hours at the Week 2, Week 6, and Month 3 Visits, is < 0 mmHg for all time points over all visits.

The study will be considered a success if both  $H_{01}$  and  $H_{02}$  are rejected.


# 8.3 Analysis Methods

All continuous study assessments will be summarized by treatment and time point (as applicable) using descriptive statistics (n, mean, median, SD, minimum, and maximum). All categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and percentages. All statistical tests will be performed at a 2-sided 5% significance level. For the IOP measurements, 2-sided tests and 2-sided 95% confidence intervals will be reported.

Mean diurnal IOP values will be constructed by averaging the three IOP measurements on each of Week 2, Week 6, and Month 3. Mean diurnal baseline IOP will be constructed as the average of the three Day 1 IOP measurements. Mean change from mean baseline diurnal IOP will be created by taking the average of the three time points on each of Week 2, Week 6, and Month 3 and subtracting the mean baseline diurnal IOP measurement.

For diurnally adjusted IOP measures, baseline will refer to the time-relevant measure at Visits 3.0 through 3.2 (e.g., IOP at 08:00 hours at Visit 3.0 will be the baseline for 08:00 hours at Visits 4.0, 5.0, and 6.0; IOP at 10:00 hours at Visit 3.1 will be the baseline for 10:00 hours at Visits 4.1, 5.1, and 6.1). For mean diurnal IOP, baseline will refer to the mean diurnal IOP at Visit 3. For all other variables, baseline is defined as the last measurement prior to the first dose of study medication. Change from baseline will be calculated as follow-up visit – baseline visit.

Percent change from diurnally adjusted baseline IOP will be determined by dividing the change from diurnally adjusted baseline by the corresponding baseline IOP value, such that a negative change from baseline will produce a negative percent change from baseline.

All primary and secondary efficacy variables, along with the planned analysis methods for those variables, are given in Table 8-1. These analyses will be performed for the ITT population for all efficacy variables and PP population for selected efficacy variables. The ITT population will be used for all efficacy subgroup analyses. Note that each subject will have one eye designated as the study eye. Only study eyes will be evaluated for all of the efficacy measures; however, both eyes will be treated. Fellow eyes will be evaluated separately for the primary analysis of the primary efficacy measure.


Table 8-1 Summary of Efficacy Variables and Analysis Methods

| | Two<br>Sample<br>T-test <sup>a</sup> | ANCOVA <sup>b</sup> | MMRM <sup>c</sup> | Fisher's<br>Exact<br>Test <sup>d</sup> | Analysis<br>Population | Missing Data<br>Imputation |
|---|---|---|---|---|---|---|
| Primary Analysis | | | | | | |
| Mean IOP at each time point at Week 2, Week 6, and Month 3 | | X | | | ITT | MCMC |
| Secondary Analyses | | | | | | |
| Mean IOP at each time point at Week 2, Week 6, and Month 3 | X | | | | ITT | MCMC |
| Month 3 | X | X | | | PP | MCMC, LOCF,<br>BOCF,<br>Observed data |
| | X | X | | | ITT | LOCF,<br>BOCF |
| | X | X | X | | ITT | Observed data |
| Mean change from diurnally adjusted baseline IOP at each post-treatment time point | X | | | | ITT | MCMC<br>LOCF,<br>Observed data |
| Mean change from baseline in diurnal IOP at each post-treatment time point | X | | | | ITT | MCMC<br>LOCF,<br>Observed data |
| Mean percent change from diurnally adjusted baseline IOP at each post-treatment time point | X | | | | ITT | Observed data |
| Percentages of subjects<br>achieving pre-specified mean,<br>mean change, and percent<br>mean change diurnal IOP<br>levels | | | | X | ITT, PP | Observed data |

<sup>&</sup>lt;sup>a</sup> Two Sample T-test comparing actual mean IOP value at each time point between PG324 and each comparator (latanoprost and Netarsudil).

# 8.3.1 Primary Efficacy Analyses

The primary analysis of the primary outcome will employ a linear model with mean IOP at the given visit (Week 2, Week 6, and Month 3) and time point (08:00, 10:00, and 16:00 hours) as the


<sup>&</sup>lt;sup>b</sup> ANCOVA model including treatment as the main effect and baseline as the covariate. Individual models will be fit for each visit and time point.

<sup>&</sup>lt;sup>c</sup> Mixed Model Repeated Measures analysis including treatment as the main effect, and baseline IOP, visit, time point, treatment\*visit, treatment\*time point, visit\*time point, and treatment\*visit\*time point as model terms. Repeated measures will be used to account for the correlation among measures within a subject. The model will include all post-dose visits and time points.

<sup>&</sup>lt;sup>d</sup> Fisher's exact test comparing the incidence in each category at each time point between PG324 and each comparator (latanoprost and Netarsudil).

response, baseline IOP as a covariate, and treatment as a main effect factor, using the intent to treat population with multiple imputation techniques (eg, Monte Carlo Markov Chain) used to impute missing data. Each time point within each visit will be modeled separately. The least squares mean differences (PG324 – comparator) between PG324 Ophthalmic Solution and each of Latanoprost Ophthalmic Solution 0.005% and Netarsudil Ophthalmic Solution 0.02% will be tested. The 2-sided p-values and associated 95% confidence intervals will be presented. For a given comparator (latanoprost and Netarsudil), if the p-value is < 0.05 and the point estimate < 0 for all time points at the Week 2, Week 6, and Month 3 Visits, then the corresponding null hypothesis will be rejected in favor of the alternative hypothesis and PG324 will be considered to be superior to the comparator.

The following SAS code will be used for multiple imputations using the Monte-Carlo Markov Chain method, where a separate model will be fit for each time point at each visit.

```
proc mi data = indata seed = 48669 out = outdata1;

mcmc initial = em;

var trt01pn baseline IOP;

run;

where
```

- *indata* is the name of the input dataset
- *outdata* is the name of the output dataset
- trt01pn is the name of the treatment group variable in numeric format
- baseline captures the baseline IOP for the given time point
- *IOP* is the name of the IOP measure.

Five complete data sets will be generated from the above code. Each complete data set will be used to analyze this primary efficacy endpoint separately using analysis of variance. Then, the SAS procedure MIANALYZE will be used to analyze the results from the 5 complete data sets to generate a combined inference. The following SAS code will be used:

```
ods output diffs = outdata2;
proc mixed data = outdata1;
class trt01pn;
model IOP=trt01pn baseline;
lsmeans trt01pn / cl pdiff;
by _Imputation_;
run;

proc sort data=outdata2;
by trt01pn _trt01pn;
run;

ods output ParameterEstimates = outdata3;
proc mianalyze data = outdata2 alpha = 0.05;
by trt01pn _trt01pn;
class trt01pn _trt01pn;
```


modeleffects *estimate*; stderr *stderr*;

run;

#### where

- *IOP* is the name of the IOP measure
- trt01pn is the name of the treatment group variable in numeric format
- *outdata2* is the name of the output dataset that contains the statistical results of the differences between treatment groups
- *outdata3* is the name of the output dataset that contains summary and inferential statistics.

## **8.3.2** Secondary Efficacy Analyses

The secondary efficacy analyses will include repeating the primary efficacy analysis on all subjects and additional analyses of the primary efficacy endpoint as well as other analyses of the secondary endpoints, as outlined below.

The primary efficacy analysis will be repeated on the ITT population using observed data only, last observation carried forward (LOCF) where LOCF will be performed using time-relevant measures; and baseline observation carried forward (BOCF) using time-relevant measures to determine the robustness of results. Additionally, the above analyses will be repeated on the PP population to determine robustness of results.

Secondary analyses of the primary endpoint will be completed using individual two-sample t-tests and 95% t-distribution confidence intervals for each comparison (PG324 vs latanoprost, PG324 vs Netarsudil at each time point (08:00, 10:00, and 16:00 at the Week 2, Week 6 and Month 3 Visits) using the ITT and PP populations. Models adjusting for baseline will only be performed on the mean IOP response variable as inference is identical between this response and the change from baseline IOP response variable in such a model based on the ITT population.

Additionally, for the mean IOP values at each time point, mixed model repeated measures will be run with baseline as the covariate; treatment, visit, time point, treatment by visit, treatment by time point, visit by time point, and treatment by visit by time point as the fixed effect factors; and subject as the random effect, repeated measure. An unstructured covariance structure will be used to model the within subject, between visit and time point variances. This allows for different variances and covariances within and between time points and visits. The treatment by visit, treatment by time point, visit by time point, and treatment by visit by time point interactions allow for a different rate of change in IOP in the different treatment arms among visits and time points. This model will be run including the Week 2, Week 6, and Month 3 visits based on the ITT population.

Percent change from diurnally adjusted baseline IOP at each time point will be analyzed using two-sample t-tests, between PG324 and each comparator, at each time point and visit, including two-sample t-tests and 95% t-distribution confidence intervals on the difference (PG324 – comparator). The analysis will be based on ITT population.


Analyses of IOP will also include summarizing the number and percentage of study eyes achieving mean diurnal IOP reduction from baseline of  $\geq 4$  to  $\geq 12$  mmHg in 2 mmHg increments and percent reduction from baseline of  $\geq 5\%$  to  $\geq 40\%$  in 5% increments at Week 2, Week 6, and Month 3. Additionally, the number and percentage of study eyes attaining a mean diurnal IOP of  $\leq 22$  to  $\leq 14$  mmHg in 1 mmHg increments will be summarized at Week 2, Week 6, and Month 3. Fisher's exact test (2-sided p-values) will be used to test the pair wise differences between treatment groups for each category at each visit. These analyses will be presented for both the ITT and PP populations with observed data only.

# 8.4 Examination of Subgroups

Subgroup analyses based upon pre-study characteristics include:

- Age: <65 years,  $\ge 65$  years
- Gender: Male, Female
- Race: Caucasian, Other
- Iris Color: Blue/Grey/Green, Brown/Black, Hazel
- Randomization stratum of baseline IOP value: <25 mmHg, ≥25 mmHg
- Maximum baseline IOP value: <23 mmHg, <25 mmHg, <27 mmHg, <30 mmHg, <32 mmHg</li>
- Prior hypotensive medication experience category 1: Combination Therapy, Prostaglandin (monotherapy), Other (monotherapy), No Prior Therapy
- Prior hypotensive medication experience category 2: Prior Prostaglandin, No Prior Prostaglandin

For each subgroup, except those defined by unmedicated baseline IOP, IOP will be compared at each post-dose time point between treatment groups (using an ANCOVA model with treatment as the main effect, baseline IOP and subgroup as covariates, and the interaction of treatment by subgroup. The least squares mean differences (test – control) between PG324 Ophthalmic Solution and each of Latanoprost Ophthalmic Solution 0.005% and Netarsudil Ophthalmic Solution 0.02% will be tested. P-values for testing the treatment difference and the interaction of treatment by subgroup will be presented. These subgroup examinations are based on the ITT population and use observed data only.

An analysis of investigative site will also be included as a subgroup analysis. The homogeneity of treatment effect across investigative sites will be examined using a similar model as the above subgroup analyses. Sites with fewer than nine subjects will be pooled together for the analysis. Results will be presented in tabular form. This analysis is based on the ITT population and use observed data only.

Statistical inference will not be made on any subgroups with fewer than nine subjects.

Subgroup analyses based upon maximum unmedicated baseline IOP in the study eye additionally will be completed for maximum baseline IOP <23 mmHg, <27 mmHg, <30 mmHg, <32 mmHg and <25 mmHg. The analysis of these IOP subgroups will be completed using only the primary endpoint analysis strategy.


## 9. SAFETY EVALUATION

# 9.1 Overview of Safety Analysis Methods

The assessment of safety and tolerability is the secondary objective of this study. All safety analyses will be carried out using the Safety Population and will include the study eye and fellow eye separately, where applicable. All tabular summaries will be provided primarily for all subjects

The assessment of safety will be evaluated by:

- Adverse events
- Comfort test (ocular tolerability)
- Heart rate and blood pressure
- Biomicroscopy of anterior segment including evaluation of cornea, conjunctiva and anterior chamber. (Fluorescein staining to be used.)
- Dilated ophthalmoscopy
- Best Corrected ETDRS Visual Acuity
- Pupil size
- Visual fields
- Pachymetry (screening only)
- IOP
- Specular microscopy
- Clinical chemistry and hematology laboratory findings

All safety variables will be descriptively summarized by treatment group at each assessment time and for relevant changes from baseline.

For complete inclusion of subjects who withdraw from the study early, the End of Study visit for safety outcomes will be defined as either Visit 6 or Early Discontinuation.

## 9.2 Extent of Exposure

Summary statistics will be presented for treatment exposure. Note that date of first dose is not collected, but will be assumed to be the Visit 3 date. Treatment exposure will be defined as the number of days that the subject was exposed to study treatment as calculated using the formula:

Treatment exposure = Date of Last Dose - Visit 3 Date + 1.

#### 9.3 Adverse Events

An adverse event is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. All AEs occurring during the study (i.e. once the subject has received one dose of study drug) will be defined as treatment emergent adverse events (TEAEs) and must be documented, regardless of the assumption of causal relationship, on the respective AE CRF. All adverse events should be documented from the time the subject receives the first dose of study drug until the subject's participation in the study has been


completed. If a subject has ongoing AEs at the time of study completion, the ongoing AEs must be followed-up and provided appropriate medical care until the event has resolved or stabilized. Documentation of AEs includes onset date, severity, action(s) taken, study medication relationship, outcome, resolution date, and seriousness.

Verbatim descriptions of AEs will be mapped to MedDRA (version: 19.0) thesaurus terms and be presented in a data listing. Treatment emergent AEs, those that occur after the first dose of study medication, will be summarized by treatment group using frequencies and proportions for each system organ class (SOC) and preferred term (PT) within each SOC. A separate summary will be presented for AEs that are related to the study drug (marked as "possibly related" or "related" in the CRF). For these summaries, Fisher's exact tests will be used to test the difference in proportions of subjects with each AE between treatment groups, SOC, and PT. Another table will be presented summarizing AEs by maximum severity. Additional summaries will be presented for serious AEs and AEs leading to test article discontinuation.

An overall summary table will be developed to report the number of events and the incidence of subjects having at least one event in the following categories:

- TEAEs
- Serious TEAEs (SAEs)
- Treatment-Related TEAEs (reported as possibly related or related to the study drug)
- Treatment-Related SAEs
- TEAEs by severity
- TEAEs leading to study drug discontinuation
- TEAEs resulting in death

While the overall summary of TEAEs will present both the number of TEAEs and the incidence of TEAEs, the other summaries will only report the incidence of TEAEs. When reporting the number of TEAEs, if the same TEAE occurs for a subject on multiple occasions the event will be counted once for each occurrence. When reporting the incidence, a subject will only be counted once if they ever experience an event within the SOC and ever experience the individual PT. Summaries will be performed using the actual treatment received.

## 9.4 Deaths, Serious Adverse Events, and Other Significant Adverse Events

An adverse event is considered "serious" if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes: Death, a life-threatening or sight-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Serious adverse events and deaths will be listed and summarized separately for the Safety population.

## 9.5 Clinical Laboratory Evaluation

Clinical laboratory results, including clinical chemistry and hematology, will be presented in data listings. Abnormal results, those above or below the normal range, will be flagged with "H" (high), "HP" (high panic), "L" (low) or "LP" (low panic) based on the laboratory ranges


provided by the lab and included in the listings. Descriptive statistics will be used to summarize continuous measures and will be presented in tabular form including change from baseline to the Month 3 visit. Shifts from baseline to the Month 3 visit will also be presented in tabular form for clinical chemistries and hematology parameters by treatment group and laboratory domain. Summary tables also will be presented for the number of subjects with abnormal values within each laboratory parameter at the end of the study. Clinical laboratory results, including clinical chemistry, hematology, and urine pregnancy test will also be listed by subject.

# 9.6 Vital Signs, Ophthalmic Exam Findings, and Other Safety Outcomes

#### 9.6.1 Vital Signs

Heart rate and blood pressure will be listed by treatment group, subject, and visit including observed values and changes from baseline. Measurements and change from baseline measurements will be summarized by treatment group and visit. Paired t-tests will be used to test within treatment group changes from baseline in vital sign parameters. Two-sided 95% CIs will be provided.

#### 9.6.2 Intraocular Pressure

Intraocular pressure will be presented in data listings. Intraocular pressure data will be summarized at each visit and time point using continuous summaries, including change from baseline, for both the study eye and the fellow eye.

# 9.6.3 Visual Acuity

Visual acuity scores will be presented in data listings. Subjects who lost three or more lines will be presented in an additional listing. Visual acuity data will be summarized at each visit using continuous summaries, including change from baseline, for both the study eye and the fellow eye. Additionally, discrete summaries of the worst change from baseline will be presented for both the study eye and the fellow eye with the following groupings based on the logMAR scores: 0 or less, >0 to +0.09, +0.10 to +0.19, +0.20 to 0.29, +0.30 or more.

#### 9.6.4 Dilated Ophthalmoscopy and Cup-to-Disc Ratio

Dilated ophthalmoscopy and cup-to-disc ratio results from Screening and Month 3 will be presented in data listings. A separate listing will be created for those subjects with a criterion change, defined as a change from "Normal" to "Abnormal" or a change from "Abnormal – Not Clinically Significant" to "Abnormal – Clinically Significant". Frequencies and percentages of normal, abnormal ophthalmoscopy results will be created for the following fields: Retina, Macula, Choroid, Optic Nerve, and Vitreous Humor. Abnormal results will further be broken down by clinical significance. A shift table of study eye and fellow eye ophthalmoscopy results will also be presented by treatment group.

Vertical cup-to-disc ratio at Screening will be summarized for the study eye and for the fellow eye by treatment group in the baseline characteristics table. Additionally, vertical cup-to-disc ratio will be summarized at follow-up visits and change from baseline to follow-up visits using


continuous summary statistics. A listing of subjects with increases of  $\geq 0.2$  in either eye at end of study will be presented.

# 9.6.5 Biomicroscopy

Biomicroscopy results will be listed for both eyes at each visit. A separate listing will be presented for subjects with a criterion change, defined as a +1 unit increase from baseline. Summaries of biomicroscopy results will also be presented for study eyes and fellow eyes by treatment group, visit, and time point in tabular form.

A summary table of the number and percentage of subjects with at least a +1 unit increase in score from baseline will be presented by region, finding, time point and eye (study eye and fellow eye). In addition to each time point, there will be summaries for "At the Final Visit" and "At Any Visit".

Additionally, for Conjunctival Hyperemia, the proportion of subjects with a one severity grade increase from baseline will be compared between Day 15 and Day 90 at each time point within a treatment arm using McNemar's test. Another summary table will be presented with the number and percentage of subjects who had a finding judged to be clinically significant by region, finding, time point and eye (study eye and fellow eye). Fisher's exact tests will be used to compare incidence between treatment groups in both tables. In addition, conjunctival hyperemia will be presented using continuous summary statistics for each visit, for the change from baseline to each post-baseline visit, and for the change from Day 15 to Day 90 visit (which will use time-specific differences [e.g. 08:00 at Day 90 – 08:00 at Day 15]). Differences between treatment groups will be tested using two-sample t-tests as well as Wilcoxon rank sum tests.

#### 9.6.6 Comfort Test (Ocular Tolerability)

Ocular discomfort after instillation of study drug will be collected at Week 2, Week 6, and Month 3, using the following categories: None, Mild, Moderate, and Severe. Discrete summaries of the discomfort categories will be provided for each visit, including the number and percentage of subjects with Moderate or Severe discomfort. Fisher's exact test will be used to compare the incidence of Moderate or Severe discomfort between treatment groups.

#### 9.6.7 Pupil Size

Pupil size (mm) will be measured at Day 1 (baseline) and Month 3 and listed for each subject. Pupil size will be summarized using continuous summary statistics for the Day 1 (baseline) and Month 3 visits as well as change from Day 1 (baseline) to Month 3 by treatment group for the study eye and fellow eye separately.

## 9.6.8 Specular Microscopy

Endothelial cell density (cells/mm2) will be measured at Day 1 (baseline) and Month 3 and listed for each subject. Endothelial cell density will be summarized using continuous summary statistics for Day 1 (baseline) and Month 3 visits as well as change from Day 1 (baseline) to Month 3 by treatment group for the study eye and fellow eye separately. Two-sample t-tests will


be used to compare treatment differences in endothelial cell density at baseline and Month 3 and change from baseline endothelial cell density to Month 3.

# 9.6.9 Visual Field Examination, Pachymetry, and Gonioscopy

Visual field examination results will be collected at Screening and Month 3 and listed for each subject. Visual field mean deviation (dB) will be summarized using continuous summary statistics for the Screening and Month 3 visits as well as change from Screening to Month 3 by treatment group for the study eye and fellow eye separately.

Central corneal thickness, collected at Screening and Month 3 will be listed for each subject. Central corneal thickness will be summarized using continuous summary statistics for the Screening and Month 3 visits as well as change from Screening to Month 3 by treatment group for the study eye and fellow eye separately. The study eye and fellow eye means at screening will also be summarized by treatment group and included with baseline characteristics.

Gonioscopy will be collected at screening for each eye and listed for each subject. Possible values will be Open Angle, Narrow Angle, and Closed Angle.


# 10. PHARMACOKINETIC EVALUATION

Not applicable.


# 11. OTHER ANALYSES

Any additional analyses conducted will be considered exploratory and enumerated in the CSR.


# 12. INTERIM ANALYSES AND DATA MONITORING

No interim analysis is planned.


# 13. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

No changes to the analyses that are planned in the protocol.


# 14. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583. (E9)

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320. (E3)


# 15. APPENDICES

**Table 15.1: Schedule of Visits and Procedures** 

| Day/Week/Month | Screen | Qual. #1 | Qual. #2<br>D1 | | | W2<br>(Day 15±3) | | W6<br>(Day 43±3) | | | M3<br>(Day 90±3) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3.0 | 3.1 | 3.2 | 4.0 | 4.1 | 4.2 | 5.0 | 5.1 | 5.2 | 6.0 | 6.1 | 6.2 |
| Hour | | 08:00 | 08:00 | 10:00 | 16:00 | 08:00 | 10:00 | 16:00 | 08:00 | 10:00 | 16:00 | 08:00 | 10:00 | 16:00 |
| Informed Consent | X | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | X | X | X | | | | | | | | | |
| Washout <sup>1</sup> | X | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | |
| Med/Ophthalmic Hist | X | X | X | | | | | | | | | | | |
| Concomitant<br>Medications | X | X | х | | | х | | | Х | | | X | | |
| HR/BP | X | X | X | | | X | | | X | | | X | | |
| Urine Pregnancy Test <sup>2</sup> | X | | | | | | | | | | | X | | |
| Clin Labs | X <sup>3</sup> | | | | | | | | | | | X | | |
| Symptoms/AEs <sup>4</sup> | X | X | X | X | X | X | X | X | X | х | X | X | Х | X |
| Comfort Test <sup>5</sup> | | | | | | X | | | X | | | X | | |
| Visual Acuity<br>(ETDRS) | X | X | х | | | X | | | X | | | X | | |
| Pupil size | | | X | | | | | | | | | X | | |
| IOP | X | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X | X | X | X | X | X | X | X | X |
| Biomicroscopy | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Specular Microscopy | X | | | | | | | | | | | X | | |
| Gonioscopy <sup>7</sup> /<br>Pachymetry <sup>8</sup> | G/P | | | | | | | | | | | P | | |
| Visual Field <sup>9</sup> | X | | | | | | | | | | | X | | |
| Ophthalmoscopy<br>(dilated) | X | | | | | | | | | | | X <sup>10</sup> | | x |
| Eye-Drop Instillation<br>Technique Evaluation | X | | | | | | | | | | | | | |
| Study Meds<br>Dispensed | | | | | X | | | X | | | X | | | |
| Collect Study Meds | | | | | | X <sup>11</sup> | | | $X^{11}$ | | | $X^{11}$ | | |
| Study Completed | | | | | | | | | | | | | | X |


Abbreviations: D, day; W, week; M, month; Med/Ophthalmic Hist, Medical/Ophthalmic History; HR/BP, heart rate/blood pressure; Clin Labs, Clinical Labs (Chemistry/Hematology); G, gonioscopy; P, pachymetry; AE, adverse event; ETDRS, early treatment diabetic retinopathy study; IOP, intraocular pressure

- 1. Subjects currently using ocular hypotensive medications must undergo a minimum washout period (Protocol Table 1 for details).
- 2. Urine pregnancy test for women of childbearing potential is required.
- 3. For subjects who are unable or unwilling to have blood drawn for clinical labs at Visit 1 (screening), the blood sample may be drawn at Visit 2 (Qualification Visit #1) so long as the results of the clinical labs are available for that subject prior to Visit 3 (Qualification Visit #2).
- 4. Ocular symptoms: Subjects will be queried at each visit "How are you feeling?" and treatment emergent AEs beginning at Visit 3 (Qualification Visit #2) will be documented on the AE form. Additional symptoms reported after screening and before randomization will be documented on the medical history form.
- 5. Comfort test: At 08:00 hour for study drug visits, subjects will be queried "Did you experience any discomfort when placing the drops in your eyes?"
- 6. Individuals returning at an unscheduled visit within 1 week are required to only remeasure IOP in both eyes (Protocol Section 7.1.2 to Section 7.1.5).
- 7. Gonioscopy evaluation up to 3 months prior to randomization is acceptable.
- 8. Pachymetry within one week of Screening is acceptable.
- 9. Entry visual field evaluation up to 3 months prior to randomization is acceptable. Visual field collection must meet the requirement for automated threshold visual field assessment (eg, 30-2 or 24-2 Humphrey) and reliability.
- 10. Ophthalmoscopy (dilated) at Visit 6.0 at 08:00 hours: this assessment should be performed for all non-completing subjects during the exit visit.
- 11. Collect used kit(s) dispensed during the previous visit. Collection of used kit(s) may occur anytime during this visit. Subjects who fail to return their used study medication as requested at their next study visit may return it at the following study visit (Protocol Section 5.11.2)


# 16. ATTACHMENTS

- PG324-CS302 Listing Shells
- PG324-CS302 Table Shells
